CLINICAL TRIAL: NCT06897462
Title: Effect of Science Research Wellness Ndo1 on Glycaemia in Adults With Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellizen Australia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEL202401
Record Dates: First submitted 2025-03-09; First posted 2025-03-27 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Prediabetes
Keywords: Diabetes; prediabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SRW Ndo1 (Experimental): Active arm
  The investigational product (IP) is a health supplement that contains 80 mg of dahlia4® (Dahlia pinnata extract), 80 mg of Eriomin® (Citrus limon extract), and 100 mg of Mulberry leaf extract (with 5% 1-deoxynojirimycin) per capsule. Excipients include Microcrystalline cellulose, Magnesium stearate, and Colloidal silicon dioxide.
  Participants will take two capsules of Ndo1 per day, before dinner, with water, for 12 weeks.
  Interventions: Dietary Supplement: SRW Ndo1

INTERVENTIONS:
Dietary Supplement: SRW Ndo1 — The investigational product (IP) is a health supplement for glycaemic control. Each capsule contains 80 mg of dahlia4® (Dahlia pinnata extract), 80 mg of Eriomin® (Citrus limon extract), and 100 mg of Mulberry leaf extract (with 5% 1-deoxynojirimycin).

SUMMARY:
The objective of this study is to test the effect of 12 weeks of supplementation SRW Ndo1 on metabolic health and general health in adults with prediabetes. The primary question it aims to answer are:

* How does SRW Ndo1 affect the Haemoglobin A1C (HbA1C) test outcome for adult individuals?
* How does SRW Ndo1 affect the body measures and blood pressures of adult individuals?

Investigators will compare the supplement to a placebo (a look-alike substance that contains no supplement) to see if SRW Ndo1 works to support normal blood sugar metabolism.

Participants will:

* Take supplement SRW Ndo1, two capsules a day for 12 weeks.
* Be asked to refrain from changing their diet and lifestyle drastically during the study and to refrain from starting new health supplements during the study.
* Visit the clinic at the start and the end of intervention for a blood test (8 hour fasting required prior to test)
* Keep a diary of their symptoms or adverse events during intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and over.
2. Prediabetes, defined as fasting plasma glucose of 6.1-6.9 mmol/L and/or HbA1c of 5.7-6.4% and/or 2 h plasma glucose of 7.8-11.0 mmol/L after ingestion of 75 g of oral glucose load. Blood tests conducted within 3 months before randomisation will be accepted.
3. Able to read and write English.
4. Has access to internet.
5. Provided informed consent to participate in the study.

Exclusion Criteria:

1. Has a medical condition known to affect the glycaemia.
2. Regular intake of a health supplement with effects on glycaemia.
3. Currently participating in another trial/study of a supplement or drug.
4. Has any known food or allergy or intolerances to the ingredients of the intervention.
5. Pregnant, trying to conceive or breastfeeding.
6. Has any current substance abuse (including tobacco, alcohol and recreational drugs) or currently in substance withdrawal.
7. Moderate to severe medical conditions (defined as a significant impact on social areas of functioning).
8. Any medical conditions that was not stable over the last 3 months.
9. Taking any prescription medication known to affect glycaemia or had a change in their medication within the last 3 months.
10. Currently taking celiprolol, metformin, or any angiotensin-converting enzyme inhibitor medications.
11. Major medical or surgical event requiring hospitalization within the last 3 months.
12. Any other medical reason that may make participation in this study pose a risk to the participant, including potential herb-drug interactions, at the discretion of the study medical supervisor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Serum Hemoglobin A1C (HbA1c) concentration | From enrollment to the end of treatment at 12 weeks
  Measured in mmol/mol. Normal range: <5.7

SECONDARY OUTCOMES:
Fasting plasma glucose concentration | From enrollment to the end of treatment at 12 weeks
  Measured in mg/dL
Weight | From enrollment to the end of treatment at 12 weeks
  Measured in kg
Body Mass Index (BMI) | From enrollment to the end of treatment at 12 weeks
  Measured in kg/m^2. Optimal range: 18.5-24.9.
Waist circumference | From enrollment to the end of treatment at 12 weeks
  Measured in cm
Blood lipids | From enrollment to the end of treatment at 12 weeks
  Total Cholesterol (TC):
  Normal: <5.2 mmol/L Borderline High: 5.2-6.2 mmol/L High: ≥6.2 mmol/L
  Triglycerides (TG):
  Normal: <1.7 mmol/L Borderline High: 1.7-2.3 mmol/L High: ≥2.3 mmol/L
  Low-Density Lipoprotein Cholesterol (LDL-C):
  Normal: <3.4 mmol/L Borderline High: 3.4-4.1 mmol/L High: ≥4.1 mmol/L
  High-Density Lipoprotein Cholesterol (HDL-C):
  Normal for Men: >1.0 mmol/L Normal for Women: >1.3 mmol/L Low: <1.0 mmol/L for Men, <1.3 mmol/L for Women
Liver functions test | From enrollment to the end of treatment at 12 weeks
  Alanine Aminotransferase (ALT):
  Normal: 0-40 U/L
  Aspartate Aminotransferase (AST):
  Normal: 0-40 U/L
  Alkaline Phosphatase (ALP):
  Normal: 40-150 U/L
  Total Bilirubin (TBIL):
  Normal: 3.4-17.1 μmol/L
  Gamma-Glutamyl Transferase (GGT):
  Normal: <60 U/L for men, <40 U/L for women
Hs-CRP test | From enrollment to the end of treatment at 12 weeks
  Measured in mg/L. Optimal: <1.0 mg/L
Systolic and diastolic blood pressure | From enrollment to the end of treatment at 12 weeks
  Measured in mmHg. Optimal range: <120/80 mmHg.
Energy questionnaire | From enrollment to the end of treatment at 12 weeks
  Measured using a 100-point Likert scale. 1 is 'extremely low energy' and 100 is 'extremely high energy'
Hunger and satiety questionnaire | From enrollment to the end of treatment at 12 weeks
  Measured using a 100-point Likert scale. 1 is 'extremely unsatisfied' and 100 is 'extremely satisfied'
Mood questionnaire | From enrollment to the end of treatment at 12 weeks
  Measured using a 100-point Likert scale. 1 is 'extremely stressed' and 100 is 'no stress at all'
Gastrointestinal symptoms questionnaire | From enrollment to the end of treatment at 12 weeks
  Measured using a 100-point Likert scale. 1 is 'No symptoms' and 100 is 'very severe symptoms'
Hypoglycemia events frequency questionnaire | From enrollment to the end of treatment at 12 weeks
  Measured using a 100-point Likert scale. 1 is 'None at all' and 100 is 'extremely high frequency'

CONTACTS AND LOCATIONS:
Locations (1):
- Baohua, Guangzhou, Guandong, China

IPD SHARING:
Plan to Share IPD: No
This is a commercial study. Due to intellectual property issues, the individual participant data will not be shared.